CLINICAL TRIAL: NCT04179851
Title: Comparison of Non-invasive to Invasive Assessment of Jugular Venous Pressure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Venovision1
Record Dates: First submitted 2019-11-21; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure; Congestion
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Thermal imaging of neck veins — Thermal imaging of neck veins

SUMMARY:
Assessment of the jugular venous pressure (JVP) is an important clinical sign and correlates with right atrial (RA) pressure. A patient with heart failure (HF) typically has an elevated JVP, but in cases of dehydration JVP may be low. Assessment of the JVP is key to the management of patients with fluid overload or needing diuretics. Currently the assessment of JVP is made by the physician by direct visualization of the neck veins. However this is inaccurate, may vary between investigators and depends largely on the patient's habitus. The JVP and RA pressures may also be directly measured by catheterization (a routine during right heart catheterization), but this is an invasive procedure that is seldom performed.

A thermal movie of the external jugular vein at a specific neck position may help to measure the JVP. In this study different modalities of JVP assessment (clinical assessment, thermal image and invasive measurement) are to be compared

Patients scheduled for right heart catheterization at the Shaare Zedek Medical Center for non-study related medical indications will be approached.

Non-invasive estimates of JVP will be performed independently prior to the right heart catheterization, during the waiting period (within 2 hours) prior to catheterization. These will include up to 2min of thermal camera recording (to be analysed offline) and a physician's JVP evaluation. The angle of the patient's upper body will be 30-60°, the rotation of the neck will be optimal for filming, and the neck area may be cooled to enhance the images. Blinding to the results will be confirmed by performance with separate investigators and separate data registration. Right heart catheterization will then be performed and RA pressure will be recorded, as well as pulmonary and wedge pressures. JVP measured by physician and thermal image will be matched with invasive catheterization (the gold standard) using Bland Altman plots and Spearmann correlation and comparison between methods will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients already scheduled for right heart catheterization for clinical indication
2. Age 18-90

Exclusion Criteria:

1. Local scar wound or bruise in the right side of the neck.
2. Current upper torso central venous catheterization such as a PICC line or dialysis catheter.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for right heart catheterization at the Shaare Zedek Medical Center for non-study related medical indications will be approached
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-02-05 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
central venous pressure (direct and indirect evaluation) | up to 30 days for analysis of the thermal images, up to 24hours for the direct measurement
  comparison of estimated venous pressure (in mmHg) to the direct measurement during right heart catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Tal Hasin, MD, Principal Investigator — SaareZMC
Locations (1):
- Shaare zedek MC, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No